CLINICAL TRIAL: NCT00532441
Title: Phase II Trial of Erlotinib in Combination With Docetaxel in Advanced Hepatocellular and Biliary Tract Carcinomas: Hoosier Oncology Group GI06-101
Brief Title: Erlotinib in Combination With Docetaxel in Advanced Hepatocellular and Biliary Tract Carcinomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Terminated due to funding issues.
Sponsor: Gabi Chiorean, MD (Other)
Collaborators: Sanofi (Industry); OSI Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Gabi Chiorean, MD, Principal Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GI06-101
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Results first posted 2016-02-12 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Erlotinib Hydrochloride; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib and Docetaxel: Biliary (Experimental): Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
  Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15
  Interventions: Drug: Erlotinib; Drug: Docetaxel
- Erlotinib and Docetaxel: Hepatocellular (Experimental): Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
  Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15
  Interventions: Drug: Erlotinib; Drug: Docetaxel

INTERVENTIONS:
Drug: Erlotinib — Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
Drug: Docetaxel — Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15

SUMMARY:
An unmet medical need exists for the successful therapy of patients with advanced hepatocellular and biliary tract malignances, with few and short lived disease responses to chemotherapy for both advanced stage hepatic and biliary carcinomas. Pre-clinical data shows cooperative antitumor activity between an epidermal growth factor receptor (EGFR) tyrosine kinase inhibitor and taxanes. The efficacy of erlotinib in combination with docetaxel will be assessed in this trial.

DETAILED DESCRIPTION:
Outline: This is a multi-center study.

Patients who meet eligibility criteria will receive treatment as follows until disease progression or excessive toxicities:

* Erlotinib 150 mg p.o. daily on days 2-7, 9-14, 16-28
* Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8, 15

Treatment cycle = 28 days

Performance Status: Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2

Life expectancy: At least 12 weeks

Hematopoietic:

* Absolute neutrophil count (ANC) > 1000 mm3
* Platelet count > 75,000 mm3
* Hemoglobin > 8 g/dL

Hepatic:

* Bilirubin < 2.0 x upper limit of normal (ULN)
* Transaminases (AST, ALT) < 5.0 x ULN if alkaline phosphatase is < 2.5 x ULN, or alkaline phosphatase < 5 x ULN if transaminases are < 1.5 x ULN.
* If not on anticoagulation: PT < 4 seconds above ULN; INR < 1.5; PTT < 1.3 x ULN.
* If on therapeutic anticoagulation, patients may have an INR > 1.5 and PTT within therapeutic range; INR will be monitored weekly until stable.
* Serum Albumin > 3.0

Renal:

* Creatinine clearance of > 60 ml/ min (by Cockcroft-Gault)

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Histological or cytological proof of hepatocellular or biliary tract carcinomas, not amenable to curative resection or transplantation.
* Prior cancer treatment completed at least 30 days prior to being registered for protocol therapy and recovered from the acute toxicity effects of the regimen.
* Patients may have had radiofrequency ablation, cryosurgery or embolization, but must have documented progressive disease with the involved lesion, or at least one previously untreated lesion.
* Patients may have had ≤ 2 prior chemotherapy regimens.
* Prior radiation therapy allowed to < 25% of the bone marrow at least 30 days prior to being registered for protocol therapy.
* Patients with biliary obstruction must have percutaneous transhepatic drainage or endoscopic stent placement prior to starting study treatment.
* Patients with a history of malignancy are eligible provided they have been curatively treated and demonstrate no evidence for recurrence of that cancer.
* Peripheral neuropathy ≤ grade 1.
* Patients must agree to abstain from frozen or fresh grapefruit or grapefruit juice for 5 days prior to, and during treatment.
* Patients must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) while on treatment and for a 12 week period thereafter.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.
* Written informed consent and HIPAA authorization for release of personal health information.
* Age ≥ 18 years at time of consent.

Exclusion Criteria:

* No previous treatment with EGFR inhibitors.
* No treatment with any investigational agent within 30 days prior to being registered for protocol therapy.
* No symptomatic brain metastasis. A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis, no longer require corticosteroids, and are asymptomatic.
* No Child-Pugh B or C liver cirrhosis.
* No active corneal erosions or history of abnormal corneal sensitivity test.
* No history of aneurysm or arteriovenous malformation.
* No hemorrhage/bleeding event > CTCAE Grade 3 within 30 days prior to begin registered for protocol therapy.
* No clinically significant infections as judged by the treating investigator.
* No condition that impairs patient's ability to swallow whole pills.
* No history of hypersensitivity to docetaxel or other drugs formulated with polysorbate 80.
* Females must not be breastfeeding.
* Patients who cannot avoid the following medications will be ineligible for the trial: midazolam, anti-mycotic agents (ketoconazole and related compounds), macrolide antibiotics (erythromycin and related compounds), nifedipine, phenobarbital, phenytoin, carbamazepine, and rifampin (induction) and anti-retrovirals (including ritonavir, saquinavir).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elena Gabriela Chiorean, M.D., Study Chair — Hoosier Oncology Group, LLC
Locations (12):
- United States (12):
  - Helen F. Graham Cancer Center, Newark, Delaware
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Rush-Presbyterian St. Luke's Medical Center, Chicago, Illinois
  - Cancer Care Center of Southern Indiana, Bloomington, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - IN Onc/Hem Associates, Indianapolis, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Medical Consultants, P.C., Muncie, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Methodist Cancer Center, Omaha, Nebraska

REFERENCES:
- [Result] Chiorean EG, Ramasubbaiah R, Yu M, Picus J, Bufill JA, Tong Y, Coleman N, Johnston EL, Currie C, Loehrer PJ. Phase II trial of erlotinib and docetaxel in advanced and refractory hepatocellular and biliary cancers: Hoosier Oncology Group GI06-101. Oncologist. 2012;17(1):13. doi: 10.1634/theoncologist.2011-0253. Epub 2011 Dec 30. PMID 22210086
- See also: Hoosier Oncology Group Home Page — http://www.hoosieroncologygroup.org

RESULTS

PARTICIPANT FLOW:
Groups:
- Hepatocellular; Biliary: erlotinib and docetaxel
Period: Overall Study
Arm/Group | Hepatocellular | Biliary
Started | 14 | 11
Completed | 13 | 11
Not Completed | 1 | 0
Not completed — Death | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Erlotinib and Docetaxel: Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
  Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15
  Erlotinib: Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
  Docetaxel: Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15
Arm/Group | Erlotinib and Docetaxel
Number analyzed (Participants) | 25
Age, Customized [Median (Full Range); unit: years]
  Age | 63.5 [41 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 15
Region of Enrollment [Number; unit: participants]
  United States | 25
ECOG Performance Status [Number; unit: participants] — ECOG Assessment Sacle:
  0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours
  4. Completely disabled; cannot carry on any selfcare; totally confined to bed or chair
  5. Dead
  participants
    ECOG 0 | 11
    ECOG 1 | 12
    ECOG 2 | 2
Cancer Type or Histologic Subtype [Number; unit: participants]
  Biliary | 11
  Hepatocellular | 14
Biliary Cancer Site [Number; unit: participants]
  Cholangiocarcoma | 6
  Gallbladder | 5
  N/A | 14
Disease Status [Number; unit: participants]
  Locally Advanced: Biliary | 0
  Locally Advanced: Hepatocellular | 4
  Metastatic: Biliary | 11
  Metastatic: Hepatocellular | 10
Previous Treatment [Number; unit: participants] — Previous treatment regimens for subjects, broken out by disease site (Biliary or Hepatocellular)
  participants
    Biliary: Chemotherapy | 7
    Biliary: Targeted therapy (sorafenib) | 0
    Biliary: Radiotherapy | 3
    Biliary: Y90 Radioembolization | 0
    Biliary: Surgery | 2
    Hepatocellular: Chemotherapy | 3
    Hepatocellular:Targeted therapy (sorafenib) | 7
    Hepatocellular:Radiotherapy | 2
    Hepatocellular: Y90 Radioembolization | 2
    Hepatocellular:Surgery | 3
Number of Prior Systemic Therapies [Number; unit: participants]
  Biliary: 1 Prior therapy | 6
  Biliary: >1 Prior Therapy | 1
  Hepatocellular: 1 Prior Therapy | 6
  Hepatocellular: >1 Prior Therapy | 2

OUTCOME MEASURES:

1. Primary Outcome: 16 Weeks Progression-free Survival
Description: To determine the rate of progression-free survival (PFS) at 16 weeks for the combination therapy of erlotinib and docetaxel for subjects in the Biliary stratum, per RECIST criteria. Progressive disease is defined as at least a 20% increase in the sum of the longest diameter of target lesions taking as reference the smallest sum recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Start of treatment until disease progression per RECIST criteria up to 16 weeks
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Biliary; Hepatocellular: Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
  Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15
  Erlotinib: Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
  Docetaxel: Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15
Arm/Group | Biliary | Hepatocellular
Number analyzed (Participants) | 11 | 14
months | 4.7 [1.6 to 6.9] | 3.5 [1.7 to 4.5]

2. Secondary Outcome: Response Rate
Description: Determine the Response Rate Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0)
Time Frame: 18 months
Measure: Number; unit: participants
Groups:
- Erlotinib and Docetaxel: Biliary; Erlotinib and Docetaxel: Hepatocellular: Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
  Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15
  Erlotinib: Erlotinib 150 mg p.o. daily, days 2-7, 9-14, 16-28
  Docetaxel: Docetaxel 30 mg/m2 IV over 30 min weekly x 3 weeks on days 1, 8 and 15
Arm/Group | Erlotinib and Docetaxel: Biliary | Erlotinib and Docetaxel: Hepatocellular
Number analyzed (Participants) | 11 | 13
participants
  Complete Response or Partial Response | 0 | 0
  Stable Disease | 7 | 6
  Progressive Disease | 4 | 7

3. Secondary Outcome: Overall Survival
Description: Determine Overall Survival
Time Frame: 18 Months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Hepatocellular | Biliary
Number analyzed (Participants) | 13 | 11
months | 6.7 [4.6 to 13.8] | 5.7 [3.6 to 21.5]

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | Erlotinib and Docetaxel
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib and Docetaxel (N=25)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 1 (1)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Investigations) | 1 (1)
DEATH NOT ASSOCIATED WITH CTCAE TERM / DEATH NOS (General disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (2)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, GI / LOWER GI NOS (Gastrointestinal disorders) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / CATHETER-RELATED (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1)
LIVER DYSFUNCTION/FAILURE (CLINICAL) (Hepatobiliary disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
PLEURAL EFFUSION (NON-MALIGNANT) (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Erlotinib and Docetaxel (N=25)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 3 (6)
ALKALINE PHOSPHATASE (Investigations) | 10 (16)
ALLERGIC REACTION/HYPERSENSITIVITY (INCLUDING DRUG FEVER) (Immune system disorders) | 1 (1)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 2 (3)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 8 (12)
ANOREXIA (Gastrointestinal disorders) | 11 (21)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 1 (1)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 8 (12)
BILIRUBIN (HYPERBILIRUBINEMIA) (Investigations) | 5 (6)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 2 (2)
CARDIAC ARRHYTHMIA - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 1 (1)
CONFUSION (Nervous system disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 10 (22)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 (12)
CREATININE (Investigations) | 1 (1)
CYTOKINE RELEASE SYNDROME/ACUTE INFUSION REACTION (Immune system disorders) | 1 (1)
DEHYDRATION (Gastrointestinal disorders) | 4 (4)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 6 (7)
DIARRHEA (Gastrointestinal disorders) | 15 (24)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 6 (11)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 7 (11)
EDEMA: LIMB (Blood and lymphatic system disorders) | 8 (10)
ESOPHAGITIS (Gastrointestinal disorders) | 1 (1)
EXTRAPYRAMIDAL/INVOLUNTARY MOVEMENT/RESTLESSNESS (Nervous system disorders) | 1 (2)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 19 (35)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 6 (9)
FISTULA, PULMONARY/UPPER RESPIRATORY / BRONCHUS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 3 (3)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 7 (13)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 11 (12)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 4 (4)
HEMOGLOBIN (Blood and lymphatic system disorders) | 6 (10)
HEMOLYSIS (E.G., IMMUNE HEMOLYTIC ANEMIA, DRUG-RELATED HEMOLYSIS) (Blood and lymphatic system disorders) | 1 (9)
HEMORRHAGE, GI / RECTUM (Gastrointestinal disorders) | 1 (1)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HEMORRHOIDS (Gastrointestinal disorders) | 2 (3)
HOT FLASHES/FLUSHES (Endocrine disorders) | 1 (1)
HYPERTENSION (Cardiac disorders) | 2 (2)
HYPOTENSION (Cardiac disorders) | 1 (1)
INCONTINENCE, ANAL (Gastrointestinal disorders) | 1 (1)
INCONTINENCE, URINARY (Renal and urinary disorders) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / LUNG (PNEUMONIA) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / UPPER AIRWAY NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INFECTION WITH UNKNOWN ANC / CONJUNCTIVA (Infections and infestations) | 1 (1)
INSOMNIA (General disorders) | 5 (5)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 4 (4)
LYMPHOPENIA (Blood and lymphatic system disorders) | 3 (3)
METABOLIC/LABORATORY - OTHER (SPECIFY, __) (Investigations) | 1 (3)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 5 (5)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 1 (1)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 8 (13)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 3 (4)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-LOWER (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 2 (2)
NAIL CHANGES (Skin and subcutaneous tissue disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 14 (22)
NEUROPATHY: SENSORY (Nervous system disorders) | 7 (9)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 2 (3)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 11 (14)
PAIN / BACK (General disorders) | 3 (5)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN / BUTTOCK (General disorders) | 1 (1)
PAIN / CHEST WALL (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / ESOPHAGUS (Gastrointestinal disorders) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 4 (5)
PAIN / GALLBLADDER (Hepatobiliary disorders) | 1 (1)
PAIN / HEAD/HEADACHE (General disorders) | 3 (4)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / LIVER (Hepatobiliary disorders) | 1 (2)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 1 (2)
PAIN / SINUS (General disorders) | 1 (1)
PAIN - OTHER (SPECIFY, __) (General disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 2 (3)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 2 (4)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 3 (4)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 9 (15)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 11 (16)
RASH: DERMATITIS ASSOCIATED WITH RADIATION / RADIATION (Skin and subcutaneous tissue disorders) | 1 (1)
RASH: HAND-FOOT SKIN REACTION (Skin and subcutaneous tissue disorders) | 2 (3)
RENAL/GENITOURINARY - OTHER (SPECIFY, __) (Renal and urinary disorders) | 1 (1)
RIGORS/CHILLS (General disorders) | 1 (1)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 2 (4)
STRICTURE/STENOSIS (INCLUDING ANASTOMOTIC), GI / DUODENUM (Gastrointestinal disorders) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / ATRIAL TACHYCARDIA/PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 1 (1)
SWEATING (DIAPHORESIS) (General disorders) | 2 (3)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 10 (15)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 9 (11)
WATERY EYE (EPIPHORA, TEARING) (Eye disorders) | 4 (4)
WEIGHT GAIN (General disorders) | 1 (2)
WEIGHT LOSS (General disorders) | 5 (6)

LIMITATIONS AND CAVEATS:
No statistical correlations with PFS and OS could be performed due to the small number of KRAS mutations.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No